CLINICAL TRIAL: NCT02379988
Title: Pilot Study For Prone Breath Hold Technique to Decrease Cardiac and Pulmonary Doses in Women Receiving Left Breast Radiotherapy
Brief Title: Prone Breath Hold Technique to Decrease Cardiac and Pulmonary Doses in Women Receiving Left Breast Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1409500149
Record Dates: First submitted 2015-01-26; First posted 2015-03-05 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Verify radiation dose to heart and lung (Experimental): Subjects will undergo the standard of care CT simulation, which includes an additional breath hold CT. Inspiratory gated breath-hold will be used. Two radiation plans will be generated: one for the CT scan performed free breathing, and one for the CT scan performed with inspiratory gated breath hold. The cardiac and lung doses will be determined. At the discretion of the treating physician, the plan with the lower cardiac and lung dose may be used to treat the patient.
  Interventions: Radiation: Verify radiation dose to heart and lung

INTERVENTIONS:
Radiation: Verify radiation dose to heart and lung — This is a pilot study to determine whether the addition of inspiratory hold (breath holding) can decrease the radiation dose that the heart and lung receives for patients being treated for left sided breast cancer.

SUMMARY:
This is a pilot study to determine whether the addition of inspiratory hold (breath holding) can decrease the radiation dose that the heart and lung receive for patients being treated for left sided breast cancer.

DETAILED DESCRIPTION:
Subjects have a standard of care CT simulation, which includes an additional breath hold CT. Inspiratory gated breath-hold will be used. Two radiation plans will be generated: one for the CT scan performed free breathing, and one for the CT scan performed with inspiratory gated breath hold. The cardiac and lung doses will be determined. At the discretion of the treating physician, the plan with the lower cardiac and lung dose may be used to treat the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Dr. Gonzalez
* ≥18 years of age
* Node-negative left breast cancer
* Invasive or DCIS breast cancer
* Prior lumpectomy
* Deemed appropriate for treatment in the prone position by the treating physician
* Able to tolerate prone position and breath hold during CT simulation

Exclusion Criteria:

* <18 years of age
* Patients requiring treatment in supine position

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-07-03 (Actual); Study Completion 2016-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor J Gonzalez, MD, Principal Investigator — University of Arizona Radiation Oncology; Uma Goyal, MD, Principal Investigator — University of Arizona Radiation Oncology
Locations (1):
- Radiation Oncology Department at the University of Arizona Heath Network, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2014 to 2016, 15 women with left-sided breast cancer were enrolled from the University of Arizona Cancer Center clinic. One was excluded from the final analysis because she did not tolerate prone positioning at the time of simulation, leaving 14 patients with evaluable pFB and pDIBH scans.
Pre-assignment Details: One patient who consented was deemed not eligible as she could not tolerate prone positioning
Period: Overall Study
Arm/Group | Verify Radiation Dose to Heart and Lung
Started | 15
Completed | 14
Not Completed | 1
Not completed — Not eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Verify Radiation Dose to Heart and Lung
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 58 [40 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Karnofsky performance status [Median (Full Range); unit: Scores on a scale] — The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
  Scores on a scale | 100 [0 to 100]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 30 [20 to 40]
Pathologic tumor stage [Count of Participants; unit: Participants] — Tumor staging was done pathologically using a combination of clinical information and pathologic examination. Tis = stage 0; T1 refers to the size and/or extent of the main tumor (higher numbers after T indicates larger tumors and/or growth into nearby tissues).
  Participants
    Tis | 4
    T1 | 10
Pathologic nodal stage [Count of Participants; unit: Participants] — Only patients with node-negative left breast cancer were eligible to participate as indicated by the pathologi nodal stage, N0. For N0 (i+), the abbreviation "i+" means that a small number of cancer cells were seen in routine stains or when a special type of staining technique, called immunohistochemistry, was used.
  Participants
    N0 | 9
    N0 (i+) | 1
    None | 4
Surgery [Count of Participants; unit: Participants]
  Conservative surgery + biopsy of sentinal node | 10
  n/a | 4
Histology [Count of Participants; unit: Participants]
  Ductal infiltrating carcinoma | 9
  Lobular infiltrating carcinoma | 1
  In-situ ductal carcinoma | 4
Tumor location [Count of Participants; unit: Participants]
  Upper Outer Quadrant (UOQ) | 6
  Upper Quadrant (UQ) | 3
  Upper Inner Quadrant (UIQ) | 2
  Lower Outer Quadrant (LOQ) | 1
  Lower Quadrant (LQ) | 2
Oncotype [Count of Participants; unit: Participants] — Number of patients where Oncotype (predict whether breast cancer will spread or come back) was assessed (yes) versus not assessed (no).
  Participants
    Yes | 5
    No | 9
Estrogen/progesterone receptors [Count of Participants; unit: Participants]
  Positive | 12
  Negative | 1
  n/a | 1
Ki67 proliferation index [Mean (Full Range); unit: Percentage of positive cells] | 16 [5 to 40]
Her2 neu immunohistochemistry [Count of Participants; unit: Participants]
  Positive | 1
  Negative | 10
  n/a | 3
Anti-hormone therapy [Count of Participants; unit: Participants]
  Yes | 11
  No | 3
Anti-her2 neu therapy [Count of Participants; unit: Participants]
  Yes | 1
  No | 13
Neoadjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 1
  No | 13
Adjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 1
  No | 13

OUTCOME MEASURES:

1. Primary Outcome: The Radiation Dose in Gy to the Heart and Lung Using Two Radiation Techniques.
Description: The primary endpoints of this study were to evaluate the feasibility of the combination of prone positioning and RPM pDIPH for breast cancer radiation treatment. Each woman enrolled in the study had 2 radiation plans generated: one for the pFB scan and one for the pDIBH scan. The mean difference between the dosimetrically determined heart, left anterior descending (LAD) artery, and left lung radiation doses were computed with the associated 95% confidence interval; however, the Wilcoxin paired signed rank test was used and listed below as the primary analysis because of the non-normal distributions.
Time Frame: Treatment Day 1 (both pFB and pDIBH scans were done on the same day)
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Verify Radiation Dose to Heart and Lung
Number analyzed (Participants) | 14
Gy
  Free breathing Heart Mean | 0.9317 (44.96)
  Breath Holding Heart mean | 0.7186 (11.43)
  Free breathing Lung mean | 0.6523 (52.78)
  Breath Holding Lung mean | 0.8746 (44.81)
  Free breathing LAD mean | 2.6159 (270.58)
  Breath holding LAD mean | 2.6231 (254.61)
Statistical Analysis 1: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — The wilcoxon paired signed rank test was used as the primary analysis because of the non-normal distributions; p = 0.0063, Wilcoxon (Mann-Whitney) — P-value for Free breathing and Breath Holding Heart Mean
Statistical Analysis 2: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — The wilcoxon paired signed rank test was used as the primary analysis because of the non-normal distributions; p = 0 .0110, Wilcoxon (Mann-Whitney) — P-value for Free breathing and Breath Holding Lung Mean
Statistical Analysis 3: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — The wilcoxon paired signed rank test was used as the primary analysis because of the non-normal distributions; p = 0.5098, Wilcoxon (Mann-Whitney) — P-value for Free breathing and Breath Holding LAD Mean

2. Secondary Outcome: Determination of Cardiac Dose and Lung Dose Reduction in Women Receiving Prone Breast Radiotherapy When Inspiratory Gating is Added.
Description: This outcome was measured by looking at the maximum dose to the heart and maximum dose to the left lung in patients using the free breathing method versus the breath holding method in the prone position. The mean of the maximum doses for each patient was taken and compared using the Wilcoxin Paired Signed Rank Test.
Time Frame: Treatment Day 1
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Verify Radiation Dose to Heart and Lung
Number analyzed (Participants) | 14
Gy
  Heart Max free breathing | 15.7029 (1424.78)
  Heart Max breath hold | 7.1869 (688.47)
  Lung max free breathing | 17.9426 (1588.08)
  Lung max breath holding | 26.6156 (1392.71)
Statistical Analysis 1: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — The wilcoxon paired signed rank test was used as the primary analysis because of the non-normal distributions; p = 0.0010, Wilcoxon (Mann-Whitney) — P-value for Heart Max Free breathing and Breath Hold
Statistical Analysis 2: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — The wilcoxon paired signed rank test was used as the primary analysis because of the non-normal distributions; p = 0.0110, Wilcoxon (Mann-Whitney) — P-value for Lung Max Free breathing and Breath Hold

3. Secondary Outcome: Heart Mean Dose Based on Breast Volume
Description: The breast volume was evaluated using the dose-volume histogram. A paired t-test was used to assess if breast volume and the mean difference for heart was statistically significant. Because paired data were generated the number of women required was less than if 2 independent samples of women were to be used.
Time Frame: Treatment Day 1
Population: The mean breast volume in the group was measured and then split into 2 groups based on breast volume, a smaller group (8), and a larger group (6). The mean breast volume was 2028.92 cc. The smaller breast volume group was less than or equal to 2028.92 cc. The larger breast volume group was >2028.92 cc.
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Verify Radiation Dose to Heart and Lung
Number analyzed (Participants) | 14
Gy
  Free breathing heart mean in smaller breast volume group: number analyzed (Participants) | 8
  Free breathing heart mean in smaller breast volume group | 109.4 (54.8)
  Breath holding heart mean in smaller breast volume group: number analyzed (Participants) | 8
  Breath holding heart mean in smaller breast volume group | 77.5 (10.4)
  Free breathing heart mean dose in larger breast volume group: number analyzed (Participants) | 6
  Free breathing heart mean dose in larger breast volume group | 71.6 (8.1)
  Breath hold heart mean dose in larger breast volume group: number analyzed (Participants) | 6
  Breath hold heart mean dose in larger breast volume group | 64.3 (8.2)
Statistical Analysis 1: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — Paired T-test; p = 0.01, Paired T-test — P-value for Large breast volume group
Statistical Analysis 2: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — Paired T-test; p = 0.10, Paired T-test — P-value for Small breast volume group

4. Secondary Outcome: Determination of Left Anterior Artery (LAD) Dose Reduction in Women Receiving Prone Breast Radiotherapy When Inspiratory Gating is Added.
Description: This outcome was measured by looking at the maximum dose to the LAD in patients using the free breathing method versus the breath holding method in the prone position. The mean of the maximum doses for each patient was taken and compared using the Wilcoxin Paired Signed Rank Test.
Time Frame: Treatment Day 1
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Verify Radiation Dose to Heart and Lung
Number analyzed (Participants) | 14
Gy
  Free breathing LAD max | 9.9154 (1166.83)
  Breath holding LAD max | 8.3896 (1108.48)
Statistical Analysis 1: Comparison: Verify Radiation Dose to Heart and Lung; Test type: Equivalence — Wilcoxon test was used due to the non-normal distribution of the data; p = 0.7776, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event collection was done through the 1 year follow-up period. It should be noted though that all adverse events recorded were in relation to the radiation therapy itself and not the study intervention of deep inspiratory breath-hold (DIBH) during prone breast RT.
Description: The intervention for this trial is a breathing technique and does not pose any risk to the patient. No adverse events were recorded in relation to the study intervention itself.
Arm/Group | Verify Radiation Dose to Heart and Lung
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT02379988/Prot_SAP_000.pdf